

Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016

Version: 1

Date: 30 MAY 2019

## STATISTICAL ANALYSIS PLAN

Protocol Number: HD-MCZ-PHII-DRF062016

Study Title: Dose-Ranging Study of the Efficacy and Safety of Miconazole Oil Used for 7

or 14 Days Compared with Vehicle in the Treatment of Otomycosis

Development Phase of Study: 2

Sponsor: Hill Dermaceuticals, Inc.

Sponsor Contact: Rosario G. Ramirez, MD

Statistical Analysis Plan based on Protocol Version: 17 April 2019/ Version 6

Statistical Analysis Plan Date: 30 May 2019

Statistical Analysis Plan Version: v1



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Authored by:

SIGNATURE: S

David Van't Hof, M.S.

Associate Manager of Statistical Programming QST Consultations, Ltd.

Reviewed by:

SIGNATURE:

Veronica Powell Chief Operating Officer QST Consultations, Ltd.

DATE: 30 My 2019

Approved by:

Rosario Ramirez

Digitally s/gned by Rosario Ramirez

DN: c=US, st=FL, l=Sanford, o=Hill Dermaceut/cals, Inc.
cn=Rosario Ramirez, email=minit\_zamirez@hillderm.com
Reason:1 am approving this document
Date: 2019.05.30 14.22.33-04'00'

SIGNATURE:

Rosario G. Ramirez, MD

Medical Director Research and Development

Hill Dermaceuticals, Inc.

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.



**Statistical Analysis Plan** Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

# TABLE OF CONTENTS

| 1. | LIST OF | ABBREVIATIONS AND DEFINITIONS OF TERMS | 5 |
|----|------------|-----------------------------------------------------|----|
| 2. | INTROD | OUCTION | 6 |
| 3. | STUDY | OBJECTIVES | 7 |
| 4. | STUDY I | DESIGN | 7 |
| 5. | EFFICA | CY AND SAFETY ENDPOINTS | 9 |
| | | eacy Endpoints | |
| | 5.1.1. | Primary Efficacy Endpoints | |
| | 5.1.2. | Secondary Efficacy Endpoints | |
| | 5.1.3. | Additional Efficacy Endpoints | |
| | 5.2. Safe | ty Endpoints | |
| 6. | STATIST | ΓΙCAL AND ANALYTICAL PLANS | 11 |
| | 6.1. Gen | eral Methodology | 11 |
| | 6.1.1. | Statistical Analysis | 11 |
| | 6.1.2. | Baseline Definition | 11 |
| | 6.1.3. | Visit Mapping | 11 |
| | 6.1.4. | Adjustments for Covariates | 12 |
| | 6.1.5. | Handling of Dropouts or Missing Data | 12 |
| | 6.1.6. | Interim Analyses and Data Monitoring | 12 |
| | 6.1.7. | Multicenter Studies | 13 |
| | 6.1.8. | Multiple Comparisons/Multiplicity | 13 |
| | 6.1.9. | Use of an Efficacy Subset of Subjects | 14 |
| | 6.1.10. | Active-Control Studies Intended to Show Equivalence | 14 |
| | 6.1.11. | Examination of Subgroups | 14 |
| | 6.2. Disp | position of Subjects | 14 |
| | 6.3. Prote | ocol Deviations | 14 |
| | 6.4. Data | Sets Analyzed | 14 |
| | 6.4.1. | Intent-to-Treat (ITT) Population | 15 |
| | 6.4.2. | Modified Intent-to-Treat (MITT) Population | 15 |
| | 6.4.3. | Per-Protocol (PP) Population | 15 |
| | 6.4.4. | Safety Population | |
| | 6.5. Dem | nographic and Other Baseline Characteristics | 16 |
| | 6.6. Prior | r and Concomitant Medications | 16 |



**Statistical Analysis Plan** Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016

Version: 1 Date: 30 MAY 2019

| | 6.7. Anal | ysis of Efficacy | |
|----|------------|--------------------------------|-----|
| | 6.7.1. | | |
| | 6.7.2. | Secondary Efficacy Analysis | |
| | 6.7.3. | Other Efficacy Analysis | .18 |
| | 6.8. Safet | ty Evaluation | |
| | 6.8.1. | Extent of Exposure | .18 |
| | 6.8.2. | Medical History | .19 |
| | 6.8.3. | Adverse Events | .19 |
| | 6.8.4. | Clinical Laboratory Evaluation | .19 |
| | 6.8.5. | Physical Examination | .19 |
| 7. | DETERM | IINATION OF SAMPLE SIZE | .19 |
| 8. | CHANGI | ES IN THE PLANNED ANALYSES | .19 |
| 9. | INDEX O | OF PLANNED TABLES | .20 |
| 10 | INDEX O | OF PLANNED LISTINGS | .80 |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

## 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE(s) adverse event(s)

ATC Anatomical Therapeutic Chemical

BID twice daily

CRF(s) case report form(s)

eCRF(s) electronic case report form(s)
FDA Food and Drug Administration

ITT intent-to-treat

LOCF last observation carried forward

MedDRA Medical Dictionary for Regulatory Activities

MIC Minimum inhibitory concentration

MITT Modified intent-to-treat number of observations

N number of subjects (sample size)

OTC over-the-counter PP per-protocol

QST QST Consultations, Ltd. SAE(s) serious adverse event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

SD standard deviation

SOP(s) Standard Operating Procedures

TEAE(s) treatment-emergent adverse event(s)

US United States

WHO World Health Organization

WHO-DDE World Health Organization Drug Dictionary



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


## 2. INTRODUCTION

Otomycosis is a fungal otitis associated with organisms from the Candida and Aspergillus genera. The signs and symptoms of otomycosis are pruritus, debris, the presence of fungal elements, and pain. While antifungal agents including miconazole are used in practice for the treatment of fungal otitis externa (also called otomycosis), there are currently no treatments approved by the United States (US) Food and Drug Administration (FDA) for this indication in humans. Miconazole is an imidazole antifungal agent that has been available by prescription and over the counter (OTC), in different formulations, for many years. It is commonly used for different types of fungal skin infections, such as Candida, ringworm, jock itch, athlete's foot, nail fungus, vaginal yeast infections, and oropharyngeal candidiasis. The purpose of this study is to gather preliminary data on the efficacy and safety of 2% miconazole oil after topical otic administration in subjects with otomycosis. The objectives of the study are to obtain preliminary evidence of the efficacy and safety of miconazole oil compared with vehicle over a 14-day treatment duration; and descriptively compare the efficacy and safety of miconazole oil over treatment durations of 7 versus 14 days. Approximately 75 male or female subjects with otomycosis will receive study drug. Subjects will be randomly assigned in a 1:1:1 ratio to receive miconazole oil [administered as 5 drops per ear at ~30 mg per drop instilled into the external ear canal of the ear(s) affected by otomycosis for 7 or 14 days, or vehicle for 14 days. Efficacy assessments will include fungal culture of the affected ear(s), assessments of clinical signs and symptoms of otomycosis, and a subject global assessment. In cases of bilateral otomycosis, both ears will be treated and evaluated by the investigator, but the ear with the worse infection at Screening/Baseline, as assessed by the investigator by taking into account both clinical signs and symptoms and fungal culture results, will be used as the study ear for efficacy analyses. If both ears are determined by the investigator to have the same degree of infection at Screening/Baseline, the left ear will be used as the study ear for the purposes of efficacy analyses.

Hill Dermaceuticals, Inc. is pursuing the development of Miconazole as a topically applied ergosterol biosynthesis inhibitor for the treatment of otomycosis. The mechanisms of action of miconazole when used topically for the treatment of fungal infections involve its actions against the fungal organisms, rather than their human host. Miconazole targets the cytochrome P450-dependent enzyme 14- $\alpha$ -sterol demethylase, an enzyme that is also involved in mammalian cholesterol synthesis, resulting in inhibition of ergosterol biosynthesis in the cell membrane.

While miconazole has not been FDA-approved for otic administration for any indication in humans, clinical studies in other countries of otically-administered miconazole have been conducted and support the efficacy of miconazole in the treatment of otomycosis. The 2% concentration of miconazole is selected for this study due to the results of an internal study



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


conducted by the sponsor *in vitro* demonstrating greater zones of inhibition against *Candida* and *Aspergillus* using the 2% concentration compared with the 1% concentration. Furthermore, the 2% miconazole concentration is commonly used for dermatophyte infections, and topical application is expected to be  $\geq$ 1000-fold the minimum inhibitory concentrations (MICs) of the *Candida* and *Aspergillus* organisms most commonly associated with human otomycosis in the US. Miconazole at a strength of 2.0% has been selected as the concentration to take forward in Phase 2 development.

This study, HD-MCZ-PHII-DRF062016, is one of the confirmatory Phase 2 trials being conducted to assess the efficacy and safety of Miconazole in subjects with otomycosis.

#### 3. STUDY OBJECTIVES

The objective of this study will be to assess the efficacy and safety of Miconazole oil compared to a placebo oil vehicle when applied twice daily (BID) for 14 days in subjects with otomycosis. Descriptively compare the efficacy and safety of miconazole oil over treatment durations of 7 versus 14 days.

#### 4. STUDY DESIGN

# 4.1. Overall Study Design

This study is a randomized, partially blinded, multiple-dose, parallel-group design study conducted at up to 10 study centers in the US. Approximately 75 male or female subjects with otomycosis will receive study drug. Subjects will be randomly assigned in a 1:1:1 ratio to receive miconazole oil [administered as 5 drops per ear at ~30 mg per drop instilled into the external ear canal of the ear(s) affected by otomycosis] for 7 or 14 days, or vehicle for 14 days. Interim assessments are planned to ensure that there is a sufficient number of subjects within each group for the primary analysis. If deemed necessary the randomization ratio may be adjusted following the interim assessments, see section 6.1.6 for details. For subjects assigned to the 14-day treatment duration with either miconazole oil or vehicle, the contents of the study drug will be blinded to both the subject and the investigator and study staff (i.e., double-blind), but the treatment duration assigned to each subject (7 or 14 days) will be unblinded to both the subject and the investigator and study staff.

At Screening/Baseline (Day 1), the subject will then begin treatment with study drug. All subjects will return to the clinic on Day 8. For subjects randomized to the 7-day treatment duration, this visit will constitute the End of Treatment Visit. Subjects randomized to the 7-day treatment duration will not administer study drug on the day of this visit. All other subjects will



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


continue to administer the study drug twice per day, up through Day 14, following the same instructions as provided at the Screening/Baseline Visit on Day 1.

All subjects will return to the clinic on Day 15. For subjects randomized to the 7-day treatment duration, this visit will constitute the Test of Cure Visit. For subjects randomized to the 14-day treatment duration, this visit will constitute the End of Treatment Visit. Subjects randomized to the 14-day treatment duration will not administer study drug on the day of this visit. Subjects randomized to the 14-day durations will return to the clinic on Day 22 for the Test of Cure Visit.

Efficacy assessments will include fungal culture of the affected ear(s), assessments of clinical signs and symptoms of otomycosis, and a subject global assessment. In cases of bilateral otomycosis, both ears will be treated and evaluated by the investigator, but the ear with the worse infection at Screening/Baseline, as assessed by the investigator by taking into account both clinical signs and symptoms and fungal culture results, will be used as the study ear for efficacy analyses. If both ears are determined by the investigator to have the same degree of infection at Screening/Baseline, the left ear will be used as the study ear for the purposes of efficacy analyses.

Safety assessments will include AEs.

## 4.1.1. Schedule of Visits and Assessments

The study schedule can be found in Section 6.1 of the protocol.

## 4.1.2. Method of Assigning Subjects to Treatment Groups

A randomization schedule will be generated in SAS® using PROC PLAN by a member in the QST Consultations, Ltd. (QST) Statistical Services department who is not associated with the conduct or analysis of the study. The randomization schedule will be stratified by site and separate lists will be produced for each site. Sites will receive sequentially numbered kits randomized in blocks of six in a 1:1:1 ratio.

At the Baseline/Day 1 visit, qualified subjects will be assigned to the lowest numerically available kit at the time of randomization. The assignment of the lowest numerically available kit number must be strictly adhered to as it is the method of randomization for this study. The kit number will be recorded in the electronic case report form (eCRF). Subjects will be randomized in a 1:1:1 ratio to one of three groups: 1) 7-day treatment with miconazole oil; 2) 14-day treatment with miconazole oil vehicle.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


# 4.1.3. Blinding

The Sponsor, the clinical research organization, the investigator, study site personnel and subjects will be blinded to the treatment assignment if the subject is randomized to a 14-day treatment group. Otherwise subjects in the 7 day treatment group will unblinded. The randomization schedule will be kept strictly confidential and accessible only to authorized persons. Only when the study has been completed, the populations determined, and the study database locked will the randomization schedule be made available for analysis.

The integrity of this clinical study must be maintained by observing the treatment blind. If an adverse event occurs which cannot be managed without knowing whether the subject is receiving active study drug or vehicle solution, the investigator should contact the unblinded sponsor staff to obtain treatment assignment information. The Medical Monitor must be notified whenever study medication is unblinded, preferably prior to unblinding a subject. The duration of treatment will not be blinded. For subjects randomized to the 14-day treatment durations, the contents of the study drug (miconazole oil versus vehicle) will be blinded. Randomized study drug will be packaged in identical bottles and will be labeled with a randomization number rather than the contents of the bottle.

For subjects randomized to the 14-day durations, if it becomes necessary to unblind a subject's treatment assignment in case of emergency, the investigator should contact the unblinded sponsor staff. A person at the sponsor organization who is not otherwise involved with the study will maintain a randomization list that will enable that person to inform the investigator of the subject's treatment allocation. The treatment allocation is to be obtained only if a medical emergency exists and knowledge of the medication being taken will influence the medical management of the subject.

#### 5. EFFICACY AND SAFETY ENDPOINTS

## 5.1. Efficacy Endpoints

The primary and secondary endpoints will be based on the investigator reporting of signs and symptoms for the study ear. Other efficacy endpoints will be based on the subject reporting of the symptom of pruritus.

# **5.1.1.** Primary Efficacy Endpoints

The primary efficacy endpoint is

• The percentage of subjects at the Test of Cure Visit with "therapeutic cure," defined as a negative mycological [fungal] culture plus "clinical cure" for the study ear. Clinical cure



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

# **5.1.2.** Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- Percentage of subjects with clinical cure at the Test of Cure Visit
- Percentage of subjects with a negative fungal culture at the Test of Cure Visit
- Percentage of subjects with a negative fungal culture at the Test of Cure visit as well as individual sign or symptom score of 0 or 1 on each of the scales for pruritus and debris and a score of 0 on each of the scales for fungal elements and pain.
- Percentage of subjects with individual signs or symptoms with a score of 0 or 1 on each of the scales for pruritus and debris and a score of 0 on each of the scales for fungal elements and pain.
- Subject global assessments at Baseline and Test of Cure as well as categorical shifts in the subject global assessment scale scores from the Screening/Baseline to the Test of Cure Visit.

Analyses may also be conducted by fungal organism isolated at Screening/Baseline if a common organism is isolated by at least 5 subjects.

## 5.1.3. Additional Efficacy Endpoints

Other efficacy endpoints based on subject reporting of pruritus will include the following:

• Subject therapeutic cure (defined as a negative mycological culture plus clinical cure) at the Test of Cure Visit for the study ear based on subject assessment of pruritus. Clinical cure is defined as the absence of all otomycosis signs and symptoms according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

## 5.2. Safety Endpoints

Safety endpoints will be the percentage of subjects with treatment-emergent AEs, with treatment-emergent defined as occurring upon or after administration of the first dose of study drug.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

#### 6. STATISTICAL AND ANALYTICAL PLANS

# 6.1. General Methodology

All statistical processing will be performed using SAS® unless otherwise stated. No interim analyses are planned.

No formal hypotheses will be tested in this study. Descriptive comparisons will be made between the micronazole oil and the oil vehicle groups for subjects randomized to the 14-day groups. Additionally, descriptive comparisons will be made between the 7-day and 14-day groups for subject's randomized to the micronazole oil treatment.

Descriptive statistics will be used to provide an overview of the efficacy and safety results. For categorical parameters, the number and percentage of subjects in each category will be presented. For continuous parameters, descriptive statistics will include n (number of subjects), mean, standard deviation (SD), median, minimum, and maximum.

The primary method of handling missing efficacy data will be the method of last observation carried forward (LOCF) imputation.

# 6.1.1. Statistical Analysis

All analyses will be performed by QST using SAS® Version 9.3 or later. All summary tables and data listings will be prepared utilizing SAS® software.

The standard operating procedures (SOPs) of QST will be followed in the creation and quality control of all data displays and analyses.

#### 6.1.2. Baseline Definition

Baseline is defined as the last non-missing assessment prior to first dose of study drug.

# 6.1.3. Visit Mapping

Data will be summarized based on nominal visit indications with the exception of data captured at early termination and unscheduled visits. Data from early termination and unscheduled visits will be summarized based on mapped visit values. The analysis windows for early termination and unscheduled visits are presented in the following table.

**Analysis Windows for Efficacy and Safety Assessments** 

| Scheduled Visit | Target Study Day | Analysis Window (Days) |
|-----------------|------------------|------------------------|
| Day 8 | 8 | 4 to 11 |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


| | | 2400.201.1111 |
|--------|----|---------------|
| Day 15 | 15 | 12 to 18 |
| Day 22 | 22 | 19 to 30 |

Data collected at early termination and unscheduled visits prior to study day 4 will not be analyzed, with the exception of those identified as baseline values. Data collected at early termination and unscheduled visits after study day 30 will not be included in the analyses.

The definition for the study day included in each analysis window is defined as below:

Study Day prior to Baseline Visit = Visit Date – Baseline Visit Date

Study Day on or after Baseline Visit = Visit Date - Baseline Visit Date + 1

If an assessment's mapped visit is a visit at which the subject has data from a scheduled visit, or if no analyses are planned for the assessment at the mapped visit, the data collected at the early termination or unscheduled visit will not be included in analyses.

In the event of multiple values from unscheduled or early termination assessments within an analysis window, the value closest to the scheduled visit target study day will be used for analyses. If two values tie as closest to the time point (for example, one value is before and the other value is after the time point), then the later value will be selected.

Data collected at all visits will be included in the data listings with visit presented as reported by the site.

## **6.1.4.** Adjustments for Covariates

Not applicable to this study.

# 6.1.5. Handling of Dropouts or Missing Data

Missing values from the Test of Cure visit from which the dichotomized Therapeutic Cure is derived will be imputed using LOCF method.

## 6.1.6. Interim Analyses and Data Monitoring

An interim assessment of the treatment allocation will be performed to ensure that there is a sufficient number of subjects within and across treatment arms. A subject's MITT status (specifically positive fungal culture at baseline) is determined only after randomization which may result in an imbalance between treatment groups. Therefore, at least one assessment during the conduct of the study is planned to ensure that there is a sufficient number of subjects within each group for the primary analysis. Once at least 10 MITT subjects have been enrolled in the 7-Day active group, the numbers of MITT subjects in the 14-Day active group and the 14-Day



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


vehicle group will be determined by an unblinded statistician; no persons involved in the day to day conduct of the study will be unblinded. Randomization allocation for future subjects may be adjusted if deemed necessary to achieve minimum number of subjects within each arm. At the time of the assessment, the 7-Day active kits will be removed from the randomization schedule for future subjects and the table below will be used as a guide for adjustments to the randomization allocation of 14-Day kits for future subjects. This assessment may be repeated in order to ascertain that a minimum enrollment of MITT subjects is met for each treatment group before study end.

| 14-Day Active | 14-Day Vehicle | Action |
|---|---|---|
| ≥ e + 3 | ≤ e − 3 | Skip 14-Day Active kits |
| ≥ e + 2 | e - 2 | Skip 14-Day Active kits with the exception of one kit at each site. One of the four lowest 14-Day Active kit numbers will be selected at random to remain in the schedule for each site. |
| e-1 to $e+2$ | e-1 to $e+2$ | No action |
| e - 2 | ≥ e + 2 | Skip 14-Day Vehicle kits with the exception of one kit at each site. One of the four lowest 14-Day Active kit numbers will be selected at random to remain in the schedule for each site. |
| ≤ e - 3 | ≥ e + 3 | Skip 14-Day Vehicle kits |

Note: e represents the expected number of subjects based on a 1:1 ratio and the current number of MITT subjects between the 14-Day active and 14-Day vehicle groups.  $e = \frac{1}{2}$  \* (Current number of MITT subjects between the 14-Day groups), non-integer results will be rounded down to the nearest integer. When determining an action the conditions of both the 14-Day Active and 14-Day Vehicle columns must be met.

## **6.1.7.** Multicenter Studies

Not applicable to this study.

## 6.1.8. Multiple Comparisons/Multiplicity

No adjustments for multiple comparisons or multiplicity will be made.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

## 6.1.9. Use of an Efficacy Subset of Subjects

Subjects with a clinical diagnosis of otomycosis confirmed by a positive fungal culture, who are randomized to study drug, have received at least one dose of study medication, and who do not have major protocol deviations will form the Per Protocol (PP) Population. The major protocol deviations will be defined at the time of evaluability evaluation, the time between the database soft lock and hard lock before unblinding.

Excluding subjects who have major protocol deviations will decrease the variability in treatment response and will allow for a better determination of dose-response relationship of miconazole.

## 6.1.10. Active-Control Studies Intended to Show Equivalence

Not applicable to this study.

## **6.1.11.** Examination of Subgroups

Not applicable to this study.

# 6.2. Disposition of Subjects

The number of subjects included in each analysis population (randomized, ITT, MITT, safety, PP) will be summarized by treatment group. The number of subjects who completed and discontinued (including the reasons for discontinuation) will be summarized for each treatment group.

The ear being treated (Left, Right, Both) will be summarized by treatment group as well as an indication of worse ear if "Both" is selected for the ear being treated.

Subjects who are excluded from an analysis population will be summarized by the reasons for exclusion based on primary reason for exclusion.

#### 6.3. Protocol Deviations

Protocol deviations will not be entered into the database. Deviations leading to exclusion from analysis populations will be identified. Protocol deviations will be presented in a by-subject listing.

## 6.4. Data Sets Analyzed

Subjects will be summarized based on the primary reason for exclusion. Below is the order to be used in summaries:



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

# 6.4.1. Intent-to-Treat (ITT) Population

All subjects who were randomized and dispensed study drug will be included in the ITT population.

# 6.4.2. Modified Intent-to-Treat (MITT) Population

All subjects in the ITT population with a clinical diagnosis of otomycosis confirmed by positive fungal culture will be included in the MITT population and analyzed according to the treatment group they were randomized. All efficacy analyses will be presented using the MITT population.

# 6.4.3. Per-Protocol (PP) Population

The PP population will be a subset of the MITT population and will include all subjects who complete the Test of Cure visit without any major protocol violations. The PP population will include subjects in the MITT population who did not meet any of the following criteria:

- Violated the inclusion/exclusion criteria
- Used an interfering concomitant medication
- Did not attend the Test of Cure visit
- Did not attend the End of Treatment visit
- Have not been compliant with the dosing regimen (i.e., subjects must have received 80%-120% of the expected applications of study medication in the study ear during participation in the study)
- Out of visit window at the Test of Cure Visit (-1/+8 days)

Subjects who discontinue from the study due to an adverse event related to study treatment, documented lack of treatment effect, or worsening of condition will be included in the PP population. Prior to breaking the blind, other additional criteria may be added to the list to accommodate for unforeseen events that occurred during the conduct of the trial that result in noteworthy study protocol violations.

All efficacy analyses will be performed on the PP population.

## 6.4.4. Safety Population

All subjects in the ITT population who received at least one dose of the study drug and had at least one post-Baseline safety assessment will be included in the safety population and analyzed



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

according to the treatment group they received. All safety analyses will be performed using the safety population.

# 6.5. Demographic and Other Baseline Characteristics

All demographic and baseline characteristic summaries will be done for the MITT, PP, and safety populations.

Sex, race, and ethnicity will be summarized by counts and percentages. Age will be summarized with descriptive statistics.

Baseline mycological culture, signs and symptoms of otomycosis, and subject global assessment will be summarized with descriptive statistics.

Medical histories will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary and presented in a by-subject listing.

## 6.6. Prior and Concomitant Medications

Concomitant medications will be coded to preferred name and Anatomical Therapeutic Chemical (ATC) classification of ingredients using the World Health Organization (WHO) Drug dictionary (WHO-DDE)

Counts and percentages will be provided to summarize the use of medications other than the study drug reported throughout the study. The number and percent of subjects who took other therapy will be shown by ATC level 2 term and preferred name. Medications which start prior to first dose will be considered prior medications. Ongoing medications and medications ending after the date of first dose will be considered concomitant medications. Medications which are both prior and concomitant will be included in both summaries. Incomplete start and end dates which could be either prior to first dose or after first dose will be considered prior to first dose.

A by-subject listing of all prior and concomitant medications will be presented.

## 6.7. Analysis of Efficacy

# 6.7.1. Primary Efficacy Analysis

The primary population for all efficacy analyses will be the MITT population. Efficacy endpoints will also be summarized for the PP population and will be considered supportive.

The percentage of subjects who demonstrate a positive outcome for each efficacy endpoint will be presented for the primary efficacy parameter as well as all secondary efficacy parameters.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


In cases of bilateral otomycosis, the ear with the worse infection at Screening/Baseline, as assessed by the investigator by taking into account both clinical signs and symptoms and fungal culture results, will be used as the study ear for efficacy analyses. If both ears are determined by the investigator to have the same degree of infection at Screening/Baseline, the left ear will be used as the study ear for the purposes of efficacy analyses.

The Test of Cure Visit is scheduled to occur on Day 15 for subjects randomized to the 7-day treatment duration, or on Day 22 for subjects randomized to the 14-day treatment durations.

The percentage of subjects with "therapeutic cure" at the Test of Cure Visit will be presented by treatment group. Subjects are defined as reaching "therapeutic cure" if they have a negative mycological culture plus "clinical cure" for the study ear, where "clinical cure" is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

In addition otomycosis signs and symptoms will be presented as the percentage of subjects with occurrences by treatment arm, assessor type (subject or investigator assessment), and visit. Subject assessments will be summarized for pruritus only.

## 6.7.2. Secondary Efficacy Analysis

The percentage of subjects with clinical cure at the Test of Cure visit will be presented by treatment group.

The same analysis will be done for the following endpoints:

- Percentage of subjects with a negative fungal culture at the Test of Cure Visit
- Percentage of subjects with a negative fungal culture at the Test of Cure visit as well as individual sign or symptom score of 0 or 1 on each of the scales for pruritus and debris and a score of 0 on each of the scales for fungal elements and pain.
- Percentage of subjects with individual signs or symptoms with a score of 0 or 1 on each of the scales for pruritus and debris and a score of 0 on each of the scales for fungal elements and pain.
- Frequency counts and percentages will be presented for the subject global assessments at Screening/Baseline and Test of Cure by treatment group. A categorical shift analysis (with categories of None, Minor, and Moderate) in the subject global assessment scale scores from the Screening/Baseline to the Test of Cure Visit will also be presented similarly. Only subjects with results at both the Screening/Baseline and the Test of Cure Visit will be considered in the shift analysis.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

In addition the subject global assessment will be presented in frequency counts and percentages for all study visits.

If feasible, analyses may also be conducted by fungal organism isolated at Screening/Baseline.

The secondary efficacy analysis will be presented on both the MITT and PP populations.

## 6.7.3. Other Efficacy Analysis

The counts and percentages of subjects with "subject therapeutic cure" at the Test of Cure Visit will be presented by treatment group. Subjects are defined as reaching "subject therapeutic cure" if they have a negative mycological culture plus "subject clinical cure" for the study ear, where "subject clinical cure" is defined as the absence of all otomycosis signs and symptoms based on subject assessed pruritus.

## **6.8. Safety Evaluation**

## **6.8.1.** Extent of Exposure

The extent of exposure to study drug in each treatment group will be summarized by total number of days of exposure, total number of applications, number of missed applications and number and percentage of subjects who are compliant. A subject will be considered compliant with the dosing regimen if the subject applied 80% to 120% of the expected number of applications while enrolled in the study.

Days of exposure = Date of last study application - Date of first study application + 1

Total Number of Applications:

2\*(Date of Last Application – Date of First Application + 1) – (Number of doses missed as collected on the case report form (CRF)) + (Number of extra doses as collected on the CRF)

Total Number of Expected Applications:

2\*(End of Treatment Visit Date – Date of Randomization).

If the total number of expected applications exceeds 14 for the 7-Day treatment group then the total number of expected applications will be set to 14. If the total number of expected applications exceeds 28 for the 14-Day treatment group then the total number of expected applications will be set to 28.

Compliance will be calculated as a percentage as 100 times the total number of applications divided by the total number of expected applications.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

# **6.8.2.** Medical History

Medical history results will only be shown in a by-subject listing.

#### 6.8.3. Adverse Events

All AEs that occur during the study will be recorded and classified on the basis of MedDRA terminology. Treatment-emergent AEs (TEAEs) are defined as AEs with an onset on or after the date of the first study drug application.

TEAEs will be summarized by treatment group, the number of subjects reporting a TEAE, system organ class, preferred name, severity, relationship to study drug (causality), and seriousness. When summarizing AEs by severity and relationship, each subject will be counted once within a system organ class or a preferred term by using the event with the highest severity and greatest relationship within each classification.

Serious AEs (SAEs) will be summarized by treatment group, severity and relationship to study drug, and individual SAEs will be listed by subject. In addition, a list of subjects who prematurely discontinue from the study due to an AE will be provided.

No statistical inference between treatments will be performed on adverse events.

Listings will be presented for all adverse events as well as for serious adverse events, and adverse events leading to discontinuation from the study.

## 6.8.4. Clinical Laboratory Evaluation

Urine pregnancy test results will only be shown in a by-subject listing.

# **6.8.5.** Physical Examination

Physical examination data will be presented in a by-subject listing.

#### 7. DETERMINATION OF SAMPLE SIZE

The sample size for this study is not based on statistical considerations and is instead intended to be a reasonable number of subjects upon which to gather preliminary information on the efficacy and safety of miconazole oil when administered via the otic route to subjects with otomycosis.

#### 8. CHANGES IN THE PLANNED ANALYSES

There are no changes in the conduct of the study or planned analyses.



**Statistical Analysis Plan** Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

# 9. INDEX OF PLANNED TABLES

| Table 14.0.1: Summary of Subject Enrollment and Evaluability | 22 |
|---|---|
| Table 14.0.2: Summary of Subjects Excluded from Analyses (Randomized Subjects) | 23 |
| Table 14.0.3: Summary of Subject Treatment Completion/Discontinuation (Randomized Subjects) | 24 |
| Table 14.1.1.1: Summary of Subject Demographics (Modified Intent-To-Treat Population) | 25 |
| Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population) | 26 |
| Table 14.1.1.3: Summary of Subject Demographics (Safety Population) | 27 |
| Table 14.1.2.1: Subject Baseline Characteristics (Modified Intent-To-Treat Population) | 28 |
| Table 14.1.2.2: Subject Baseline Characteristics (Per-Protocol Population) | 30 |
| Table 14.1.2.3: Subject Baseline Characteristics (Safety Population) | 32 |
| Table 14.2.1.1: Summary of Primary Efficacy Endpoint: Therapeutic Cure at Test of Cure (Modified Intent-to-Treat Population) | 34 |
| Table 14.2.1.2: Summary of Primary Efficacy Endpoint: Therapeutic Cure at Test of Cure (Protocol Population) | |
| Table 14.2.2.1.1: Summary of Secondary Efficacy Endpoints: Mycological Culture and Individual Signs and Symptoms (Modified Intent-to-Treat Population) | 36 |
| Table 14.2.2.1.2: Summary of Secondary Efficacy Endpoints: Mycological Culture and Individual Signs and Symptoms Endpoints (Per-Protocol Population | n) 37 |
| Table 14.2.2.2.1: Summary of Secondary Efficacy Endpoint: Subject Global Assessment (Modified Intent-to-Treat Population) | 38 |
| Table 14.2.2.2.2: Summary of Secondary Efficacy Endpoint: Subject Global Assessment (Per<br>Protocol Population) | |
| Table 14.2.2.3.1: Otomycosis Mycological Culture Through Time (Modified Intent-To-<br>Treat Population) | 40 |
| Table 14.2.2.3.2: Otomycosis Mycological Culture Through Time (Per-Protocol Population). | 41 |
| Table 14.2.2.4.1: Investigator Assessed Pruritus Through Time (Modified Intent-To-<br>Treat Population) | 42 |
| Table 14.2.2.4.2: Investigator Assessed Pruritus Through Time (Per-Protocol Population) | 44 |
| Table 14.2.2.5.1: Debris Through Time (Modified Intent-To-Treat Population) | 46 |
| Table 14.2.2.5.2: Debris Through Time (Per-Protocol Population) | 48 |
| Table 14.2.2.6.1: Presence of Fungal Elements Through Time (Modified Intent-To-<br>Treat Population) | 50 |



| Sta | tisti | cal | Ana | lvsis | Plar |
|-----|-------|-----|-----|-------|------|

Statistical Analysis Plan Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016

| V CISIOII. I |
|-------------------|
| Date: 30 MAY 2019 |

| Date: 30 MAY 201 | 9 |
|---|---|
| Table 14.2.2.6.2: Presence of Fungal Elements Through Time (Per-Protocol Population)5 | 1 |
| Table 14.2.2.7.1: Pain Through Time (Modified Intent-to-Treat Population) | 2 |
| Table 14.2.2.7.2: Pain Through Time (Per-Protocol Population)5 | 3 |
| Table 14.2.2.8.1: Subject Global Assessment Through Time (Modified Intent-To-<br>Treat Population) | 4 |
| Table 14.2.2.8.2: Subject Global Assessment Through Time (Per-Protocol Population)5 | 5 |
| Table 14.2.3.1.1: Summary of Other Efficacy Endpoint: Subject Therapeutic Cure at Test of Cure (Modified Intent-to-Treat Population) | 6 |
| Table 14.2.3.1.2: Summary of Other Efficacy Endpoint: Subject Therapeutic Cure at Test of Cure (Per-Protocol Population) | 7 |
| Table 14.2.3.2.1: Subject Assessed Pruritus Through Time (Modified Intent-To-<br>Treat Population) | 8 |
| Table 14.2.3.2.2: Subject Assessed Pruritus Through Time (Per-Protocol Population)6 | 0 |
| Table 14.3.1.1: Summary of Extent of Exposure (Modified Intent-To-Treat Population)6 | 2 |
| Table 14.3.1.2: Summary of Extent of Exposure (Per-Protocol Population) | 3 |
| Table 14.3.1.3: Summary of Extent of Exposure (Safety Population) | 4 |
| Table 14.3.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) | 5 |
| Table 14.3.2.2: Summary of Treatment-Emergent Adverse Events Leading to Permanent Withdrawal of Study Drug and/or Early Discontinuation From Study (Safety Population) | 9 |
| Table 14.3.2.3: Summary of Treatment-Emergent Adverse Events (Safety Population) | 0 |
| Table 14.3.2.4: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population) | 1 |
| Table 14.3.2.5: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug (Safety Population) | |
| Table 14.3.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) | |
| Table 14.3.3.2: Summary of Treatment-Emergent Serious Adverse Events (Safety Population).7 | 7 |
| Table 14.3.3.3: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population) | 8 |
| Table 14.3.3.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship to Study Drug (Safety Population) | 9 |



**Statistical Analysis Plan** Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.0.1: Summary of Subject Enrollment and Evaluability

| | 7-Day Miconazole Oil | 14-Day Miconazole Oil | 14-Day Vehicle Oil |
|---|---|---|---|
| Number of Subjects Randomized | XX | XX | XX |
| Number of Subjects Excluded from the ITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included in the ITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the MITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included in the MITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included in the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included in the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



**Statistical Analysis Plan** Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.0.2: Summary of Subjects Excluded from Analyses (Randomized Subjects)

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Number of Subjects Excluded from the ITT Population Reason for Exclusion from the ITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Dispensed Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the MITT Population Reason for Exclusion from the MITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Dispensed Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Positive Otomycosis Diagnosis | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the Safety Population<br>Reason for Exclusion from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Dispensed Study Drug | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| No Post Baseline Assessment | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the PP Population<br>Reason for Exclusion from the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Dispensed Study Drug | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| No Positive Otomycosis Diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Violated the inclusion/exclusion criteria | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Used an interfering concomitant medication | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Did not attend the Test of Cure Visit | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Have not been compliant with the dosing regimen | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Out of visit window at the Test of Cure Visit | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.0.3: Summary of Subject Treatment Completion/Discontinuation (Randomized Subjects)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Completed Study | , | , , | , , , |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation | | | |
| Adverse Event | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost To Follow-Up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pregnancy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Protocol Deviation | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Withdrawal by Subject | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Withdrawal by Parent/Guardian | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Physician Decision | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Study Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other <sup>a</sup> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.1.2 for other discontinuation reasons.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.1.1: Summary of Subject Demographics (Modified Intent-To-Treat Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Age (years) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| n | XX | XX | XX |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Female | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Ethnicity | | | |
| n | XX | XX | XX |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Race | | | |
| n | XX | XX | XX |
| American Indian or Alaska Native | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Other <sup>a</sup> | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.4.1 for a complete list of all other races.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Age (years) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| n | XX | XX | XX |
| Male | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Female | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Ethnicity | | | |
| n | XX | XX | XX |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Race | | | |
| n | XX | XX | XX |
| American Indian or Alaska Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Asian | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Black or African American | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| White | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other <sup>a</sup> | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.4.1 for a complete list of all other races.

 $SOURCE: USERNAME \verb|\SPONSOR| PROJECT \verb|\JOBNAME| (DATE, TIME)$ 



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.1.3: Summary of Subject Demographics (Safety Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Age (years) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| n | XX | XX | XX |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Female | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Ethnicity | | | |
| n | XX | XX | XX |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Race | | | |
| n | XX | XX | XX |
| American Indian or Alaska Native | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| White | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Other <sup>a</sup> | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.4.1 for a complete list of all other races.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.2.1: Subject Baseline Characteristics (Modified Intent-To-Treat Population) 

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Otomycosis Mycological Culture | | | |
| n | XX | XX | XX |
| Positive | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pruritus | | | |
| Subject Assessed | | | |
| n | XX | XX | XX |
| None | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Investigator Assessed | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Table only includes assessments of the study ear.

 $SOURCE: USERNAME \verb|SPONSOR|| PROJECT \verb|JOBNAME|| (DATE, TIME)$ 



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.1.2.1: Subject Baseline Characteristics (Modified Intent-To-Treat Population) 

| | 7-Day Miconazole Oil | 14-Day Miconazole Oil | 14-Day Vehicle Oil |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Debris | | · | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scant | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Heavy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Presence of Fungal Elements | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | XX (XX.X%) | XX (XX.X%) |
| Pain | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Subject Global Assessment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Minor | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Table only includes assessments of the study ear.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.2.2: Subject Baseline Characteristics (Per-Protocol Population)


| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Otomycosis Mycological Culture | <del>.</del> | | |
| n | XX | XX | XX |
| Positive | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pruritus | | | |
| Subject Assessed | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Investigator Assessed | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Table only includes assessments of the study ear.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.2.2: Subject Baseline Characteristics (Per-Protocol Population) 

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Debris | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scant | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Presence of Fungal Elements | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Subject Global Assessment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Minor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Table only includes assessments of the study ear.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.2.3: Subject Baseline Characteristics (Safety Population) 

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Otomycosis Mycological Culture | | | |
| n | XX | XX | XX |
| Positive | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pruritus | | | |
| Subject Assessed | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Investigator Assessed | | | |
| n | XX | XX | XX |
| None | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | $xx(x_0,x_0)$ | xx ( xx.x%) |

Note: Table only includes assessments of the study ear.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.1.2.3: Subject Baseline Characteristics (Safety Population) 

| | 7-Day Miconazole Oil | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Debris | (N=xx) | (N-XX) | (IN=XX) |
| n<br>N | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scant | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Presence of Fungal Elements | | | |
| n | XX | XX | XX |
| Absent | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Present | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Pain | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Subject Global Assessment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Minor | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | XX (XX.X/0)<br>XX (XX.X%) | xx ( xx.x%) | XX (XX.X%) |

Note: Table only includes assessments of the study ear.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.1.1: Summary of Primary Efficacy Endpoint: Therapeutic Cure at Test of Cure (Modified Intent-to-Treat Population)

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Therapeutic Cure <sup>a</sup> at Test of Cure | . , | | |
| Achieved | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Therapeutic Cure is defined as a negative mycological culture plus Clinical Cure for the study ear. Clinical Cure is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

Note: Last observation carried forward (LOCF) used to impute missing values.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.1.2: Summary of Primary Efficacy Endpoint: Therapeutic Cure at Test of Cure (Per-Protocol Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Therapeutic Cure <sup>a</sup> at Test of Cure | | | |
| Achieved | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Not Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Therapeutic Cure is defined as a negative mycological culture plus Clinical Cure for the study ear. Clinical Cure is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

Note: Last observation carried forward (LOCF) used to impute missing values.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.1.1: Summary of Secondary Efficacy Endpoints: Mycological Culture and Individual Signs and Symptoms (Modified Intent-to-Treat Population)

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Clinical Cure a at Test of Cure | , | <u> </u> | , |
| Achieved | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Achieved | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| legative Mycological Culture at Test of Cure | | | |
| Achieved | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Achieved | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| legative Mycological Culture and Individual Sign or | | | |
| ymptom Score of 0 or 1 on each of the Scales for Pruritus | | | |
| nd Debris and a Score of 0 on each of the Scales for Fungal | | | |
| lements and Pain at Test of Cure. | | | |
| Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ndividual Sign or Symptom Score of 0 or 1 on each of the | | | |
| cales for Pruritus and Debris and a Score of 0 on each of the | | | |
| cales for Fungal Elements and Pain at Test of Cure. | | | |
| Achieved | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

 <sup>&</sup>lt;sup>a</sup> Clinical Cure is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.
 Note: Last observation carried forward (LOCF) used to impute missing values.


Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.1.2: Summary of Secondary Efficacy Endpoints: Mycological Culture and Individual Signs and Symptoms Endpoints (Per-Protocol Population)

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Clinical Cure a at Test of Cure | | | |
| Achieved | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Achieved | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| legative Mycological Culture at Test of Cure | | | |
| Achieved | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Achieved | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Negative Mycological Culture and Individual Sign or | | | |
| ymptom Score of 0 or 1 on each of the Scales for Pruritus | | | |
| nd Debris and a Score of 0 on each of the Scales for Fungal | | | |
| lements and Pain at Test of Cure. | | | |
| Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ndividual Sign or Symptom Score of 0 or 1 on each of the | | | |
| cales for Pruritus and Debris and a Score of 0 on each of the cales for Fungal Elements and Pain at Test of Cure. | | | |
| Achieved | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Not Achieved | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Clinical Cure is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

Note: Last observation carried forward used to impute missing values.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.2.1: Summary of Secondary Efficacy Endpoint: Subject Global Assessment (Modified Intent-to-Treat Population)

| Subject Global Assessment | 7-Day Miconazole Oil (N=xx) Baseline Test of Cure | 14-Day Miconazole Oil (N=xx) Baseline Test of Cure | 14-Day Vehicle Oil (N=xx) Baseline Test of Cure |
|---|---|---|---|
| n | XX XX | XX XX | XX XX |
| None | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) |
| Minor | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) | xx(xx.x%) $xx(xx.x%)$ |
| Moderate | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) |
| | Test of Cure | Test of Cure | Test of Cure |
| Baseline | None Minor Moderate | None Minor Moderate | None Minor Moderate |
| None | xx(xx.x%) xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) xx(xx.x%) x | xx(xx.x%) xx(xx.x%) xx(xx.x%) |
| Minor | XX(XX.X%) $XX(XX.X%)$ $XX(XX.X%)$ | xx(xx.x%) $xx(xx.x%)$ $xx(xx.x%)$ | xx(xx.x%) xx(xx.x%) xx(xx.x%) |
| Moderate | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) x | xx(xx.x%) $xx(xx.x%)$ $xx(xx.x%)$ |

Note: No imputation of missing values.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.2: Summary of Secondary Efficacy Endpoint: Subject Global Assessment (Per-Protocol Population)

| Subject Global Assessment | 7-Day Miconazole Oil (N=xx) Baseline Test of Cure | 14-Day Miconazole Oil (N=xx) Baseline Test of Cure | 14-Day Vehicle Oil (N=xx) Baseline Test of Cure |
|---|---|---|---|
| n | XX XX | XX XX | XX XX |
| None | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) |
| Minor | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) | xx(xx.x%) $xx(xx.x%)$ |
| Moderate | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) |
| | Test of Cure | Test of Cure | Test of Cure |
| Baseline | None Minor Moderate | None Minor Moderate | None Minor Moderate |
| None | xx(xx.x%) xx(xx.x%) xx(xx.x%) | xx(xx.x%) xx(xx.x%) xx(xx.x%) x | xx(xx.x%) xx(xx.x%) xx(xx.x%) |
| Minor | XX(XX.X%) $XX(XX.X%)$ $XX(XX.X%)$ | xx(xx.x%) $xx(xx.x%)$ $xx(xx.x%)$ | xx(xx.x%) xx(xx.x%) xx(xx.x%) |
| Moderate | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) x | xx(xx.x%) $xx(xx.x%)$ $xx(xx.x%)$ |

Note: No imputation of missing values.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.3.1: Otomycosis Mycological Culture Through Time (Modified Intent-To-Treat Population)

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| tomycosis Mycological Culture<br>Baseline | | | |
| n | XX | XX | XX |
| Positive | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| Positive | | xx (xx.x%) | xx (xx.x%) |
| Negative | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| Positive | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Negative | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.3.2: Otomycosis Mycological Culture Through Time (Per-Protocol Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| tomycosis Mycological Culture | , , | , , | ` ' |
| Baseline | | | |
| n | XX | XX | XX |
| Positive | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| Positive | | xx (xx.x%) | xx ( xx.x%) |
| Negative | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| Positive | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| Positive | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Negative | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.4.1: Investigator Assessed Pruritus Through Time (Modified Intent-To-Treat Population)


| | 7-Day Miconazole Oil | 14-Day Miconazole Oil | 14-Day Vehicle Oil |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Investigator Assessed Pruritus | | | |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx ( xx.x%) |
| Mild | | xx (xx.x%) | xx ( xx.x%) |
| Moderate | | xx ( xx.x%) | xx ( xx.x%) |
| Severe | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.4.1: Investigator Assessed Pruritus Through Time (Modified Intent-To-Treat Population) 

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| nvestigator Pruritus | | | |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | XX (XX.X%) | xx (xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.4.2: Investigator Assessed Pruritus Through Time (Per-Protocol Population)


| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Investigator Assessed Pruritus | | | |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx (xx.x%) |
| Mild | | xx (xx.x%) | xx ( xx.x%) |
| Moderate | | xx (xx.x%) | xx ( xx.x%) |
| Severe | | xx ( xx.x%) | xx (xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | $XX (XX.X^{0})$ | xx (xx.x%) | xx (xx.x%) |
| Mild | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.4.2: Investigator Assessed Pruritus Through Time (Per-Protocol Population)


| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| nvestigator Pruritus | | | |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.5.1: Debris Through Time

(Modified Intent-To-Treat Population) 

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Debris | | | |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scant | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx (xx.x%) |
| Scant | | xx (xx.x%) | xx ( xx.x%) |
| Moderate | | xx (xx.x%) | xx (xx.x%) |
| Heavy | | xx (xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Scant | XX (XX.X%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.5.1: Debris Through Time (Modified Intent-To-Treat Population) 

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Debris | | | |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scant | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.5.2: Debris Through Time (Per-Protocol Population) 

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Debris | | | |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scant | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx (xx.x%) |
| Scant | | xx ( xx.x%) | xx (xx.x%) |
| Moderate | | xx (xx.x%) | xx (xx.x%) |
| Heavy | | xx ( xx.x%) | xx (xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Scant | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Heavy | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.5.2: Debris Through Time (Per-Protocol Population) 

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Pebris | | | |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scant | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Heavy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.6.1: Presence of Fungal Elements Through Time (Modified Intent-To-Treat Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Presence of Fungal Elements<br>Baseline | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| Absent | | xx ( xx.x%) | xx ( xx.x%) |
| Present | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.6.2: Presence of Fungal Elements Through Time (Per-Protocol Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Presence of Fungal Elements<br>Baseline | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| Absent | | xx ( xx.x%) | xx ( xx.x%) |
| Present | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.7.1: Pain Through Time (Modified Intent-to-Treat Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Pain | | | |
| Baseline | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| Absent | | xx (xx.x%) | xx ( xx.x%) |
| Present | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| Absent | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.7.2: Pain Through Time (Per-Protocol Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Pain | | | |
| Baseline | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| Absent | | xx (xx.x%) | xx ( xx.x%) |
| Present | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Present | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| Absent | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Present | xx (xx.x%) | xx (xx.x%) | $XX \left( XX.X\% \right)$ |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.2.8.1: Subject Global Assessment Through Time (Modified Intent-To-Treat Population)

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Subject Global Assessment | (IV AA) | (14 AA) | (11 AA) |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Minor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx (xx.x%) |
| Minor | | xx (xx.x%) | xx (xx.x%) |
| Moderate | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Minor | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Minor | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.2.8.2: Subject Global Assessment Through Time (Per-Protocol Population)

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| ubject Global Assessment | | · | |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Minor | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx (xx.x%) |
| Minor | | xx (xx.x%) | xx ( xx.x%) |
| Moderate | | xx ( xx.x%) | xx (xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Minor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Minor | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.3.1.1: Summary of Other Efficacy Endpoint: Subject Therapeutic Cure at Test of Cure (Modified Intent-to-Treat Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Subject Therapeutic Cure <sup>a</sup> at Test of Cure | | | |
| Achieved | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Therapeutic Cure is defined as a negative mycological culture plus Clinical Cure based on subject assessment of pruritus for the study ear. Clinical Cure is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

Note: Last observation carried forward used to impute missing values.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.2.3.1.2: Summary of Other Efficacy Endpoint: Subject Therapeutic Cure at Test of Cure (Per-Protocol Population)

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Subject Therapeutic Cure <sup>a</sup> at Test of Cure | | | |
| Achieved | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Achieved | XX ( XX.X%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Therapeutic Cure is defined as a negative mycological culture plus Clinical Cure based on subject assessment of pruritus for the study ear. Clinical Cure is defined as the absence of all otomycosis signs and symptoms based on Investigator assessment according to the scales for each individual sign or symptom and with absence defined as a score of 0 on each of the scales for pruritus, debris, fungal elements, and pain.

Note: Last observation carried forward used to impute missing values.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.3.2.1: Subject Assessed Pruritus Through Time (Modified Intent-To-Treat Population)


| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Subject Assessed Pruritus | | | |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx (xx.x%) |
| Mild | | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | | xx ( xx.x%) | xx ( xx.x%) |
| Severe | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.3.2.1: Subject Assessed Pruritus Through Time (Modified Intent-To-Treat Population) 

| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Subject Assessed Pruritus (cont.) | | | |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.3.2.2: Subject Assessed Pruritus Through Time (Per-Protocol Population)


| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Subject Assessed Pruritus | · | · | |
| Baseline | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Mild | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| On Treatment | | | |
| n | NA | XX | XX |
| None | | xx (xx.x%) | xx (xx.x%) |
| Mild | | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | | xx (xx.x%) | xx ( xx.x%) |
| Severe | | xx ( xx.x%) | xx ( xx.x%) |
| End of Treatment | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.2.3.2.2: Subject Assessed Pruritus Through Time (Per-Protocol Population)


| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| bject Assessed Pruritus (cont.) | | · | |
| Test of Cure | | | |
| n | XX | XX | XX |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Subjects in the 14-day treatment duration will have the follow-up visit schedule On Treatment – Day 8, End of Treatment – Day 15, and Test of Cure – Day 22. Subjects in the 7-day treatment durations will have the follow-up visit schedule End of Treatment – Day 8, and Test of Cure – Day 15.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.3.1.1: Summary of Extent of Exposure (Modified Intent-To-Treat Population)

| 7-Day Miconazole Oil (N=xx) | Total Amount of<br>Study Drug Used (g) | Total Number of<br>Days of Exposure | Total Number of Applications | Total Number of Missed Applications | | Compliant <sup>a</sup> |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | Yes | xx ( xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( xx.x%) |
| SD | XX.X | XX,X | XX.X | XX.X | | ( ' ' ' ' ' ' ' |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | |
| 14-Day Miconazole Oil (N=xx) | | | | | | |
| n | XX | XX | XX | XX | Yes | xx (xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | |
| 14-Day Vehicle Oil (N=xx) | | | | | | |
| n | xx | XX | XX | XX | Yes | xx (xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | |

<sup>&</sup>lt;sup>a</sup> A subject was considered compliant with the dosing regimen if the subject applied at least 80% but no more than 120% of the expected applications while enrolled in the study.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.3.1.2: Summary of Extent of Exposure (Per-Protocol Population)

| | Total Amount of<br>Study Drug Used (g) | Total Number of<br>Days of Exposure | Total Number of Applications | Total Number of Missed Applications | | Comp | olianta |
|---|---|---|---|---|---|---|---|
| 7-Day Miconazole Oil (N=xx) | | | | | | | |
| n | XX | XX | XX | XX | Yes | xx ( | xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( | xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | | |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | | |
| 14-Day Miconazole Oil (N=xx) | | | | | | | |
| n | XX | XX | XX | XX | Yes | xx ( | xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( | xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | | |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | | |
| 14-Day Vehicle Oil (N=xx) | | | | | | | |
| n | XX | XX | XX | XX | Yes | xx ( | xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( | xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | ` | ĺ |
| Median | XX.XX | XX.XX | XX,XX | XX.XX | | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | | |

<sup>&</sup>lt;sup>a</sup> A subject was considered compliant with the dosing regimen if the subject applied at least 80% but no more than 120% of the expected applications while enrolled in the study.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.3.1.3: Summary of Extent of Exposure (Safety Population)

| | Total Amount of<br>Study Drug Used (g) | Total Number of<br>Days of Exposure | Total Number of Applications | Total Number of<br>Missed Applications | | Comp | olianta |
|---|---|---|---|---|---|---|---|
| 7-Day Miconazole Oil (N=xx) | | | | | | | |
| n | XX | XX | XX | XX | Yes | xx ( | xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( | xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | | |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | | |
| 14-Day Miconazole Oil (N=xx) | | | | | | | |
| n | XX | XX | XX | XX | Yes | xx ( | xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( | xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | | |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | | |
| 14-Day Vehicle Oil (N=xx) | | | | | | | |
| n | XX | XX | XX | XX | Yes | xx ( | xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | No | xx ( | xx.x%) |
| SD | XX.X | XX.X | XX.X | XX.X | | | ŕ |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | | | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | | | |

<sup>&</sup>lt;sup>a</sup> A subject was considered compliant with the dosing regimen if the subject applied at least 80% but no more than 120% of the expected applications while enrolled in the study.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| <u>-</u> | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Number (%) of Subjects Reporting At Least One Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects Reporting At Least One Serious Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Discontinued Study Drug due to Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| By Subject<br>Maximum Severity | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Strongest Relationship to Study Drug | | | |
| Not Suspected | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

 $SOURCE: USERNAME \verb|SPONSOR|| PROJECT \verb|JOBNAME|| (DATE, TIME)$ 



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| y Subject | | · | |
| Maximum Severity within Relationship to Study Drug | | | |
| Not Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Number Events Reported | XX | xx | XX |
| By Event | | | |
| Serious | | | |
| No | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Death | | | |
| No | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Discontinuation of Study Drug | | | |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| | AA ( AA.A/v) | AA ( AA.A/0) | AA ( AA.A/0) |
| Severity | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | XX (XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Relationship to Study Drug | | | |
| Not Suspected | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Suspected | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| By Event | | | |
| Severity within Relationship to Study Drug | | | |
| Not Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.2.2: Summary of Treatment-Emergent Adverse Events Leading to Permanent Withdrawal of Study Drug and/or Early Discontinuation From Study (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

Note: MedDRA dictionary (Version 20.1)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

# Table 14.3.2.3: Summary of Treatment-Emergent Adverse Events (Safety Population) (Page 1 of xx)

| System Organ Class <sup>a</sup> Preferred Term | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

Note: MedDRA dictionary (Version 20.1)

 $SOURCE: USERNAME \verb|SPONSOR|| PROJECT \verb|JOBNAME|| (DATE, TIME)$ 

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.2.4: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | <u>Severity</u> | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|---|
| System Organ Class | Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

Note: MedDRA dictionary (Version 20.1)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.2.5: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | Relationship | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|---|
| System Organ Class | Not Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Not Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

Note: MedDRA dictionary (Version 20.1)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the strongest reported relationship.


Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| _ | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| Number (%) of Subjects Reporting At Least One Serious Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Discontinued Study Drug due to Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| By Subject Maximum Severity Mild Moderate Severe | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| Strongest Relationship to Study Drug<br>Not Suspected<br>Suspected | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

 $SOURCE: USERNAME \verb|SPONSOR|| PROJECT \verb|JOBNAME|| (DATE, TIME)$ 



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil (N=xx) |
|---|---|---|---|
| By Subject | | | |
| Maximum Severity within Relationship to Study Drug | | | |
| Not Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019
Table 14.3.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics

(Safety Population) 

| | 7-Day Miconazole Oil (N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Number of Serious Events Reported | xx | xx | xx |
| By Event | | | |
| Death | | | |
| No | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Yes | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinuation of Study Drug | | | |
| No | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severity | | | |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | XX (XX.X%) | xx(xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Relationship to Study Drug | | | |
| Not Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: 30 MAY 2019

Table 14.3.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| Severity within Relationship to Study Drug | | | |
| By Event | | | |
| Not Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Suspected | | | |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.3.3.2: Summary of Treatment-Emergent Serious Adverse Events (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil (N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|
| System Organ Class | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

Note: MedDRA dictionary (Version 20.1)

 $SOURCE: USERNAME \verb|SPONSOR|| PROJECT \verb|JOBNAME|| (DATE, TIME)$ 

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.3.3.3: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population)

System Organ Class<sup>a</sup> 7-Day Miconazole Oil 14-Day Miconazole Oil 14-Day Vehicle Oil Preferred Term Severity (N=xx)(N=xx)(N=xx)System Organ Class Mild xx (xx.x%)xx.x%xx (xx.x%)Moderate xx.x%xx (xx.x%)xx ( xx (xx.x%)Severe xx (xx.x%)xx (xx.x%)xx (xx.x%)Preferred Term Mild xx.x%xx (xx.x%)xx (xx.x%)Moderate xx (xx.x%)xx (xx.x%)xx ( xx.x%xx ( xx.x%) Severe xx (xx.x%)xx (xx.x%)

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

Note: MedDRA dictionary (Version 20.1)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Table 14.3.3.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship to Study Drug (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Relationship | 7-Day Miconazole Oil<br>(N=xx) | 14-Day Miconazole Oil<br>(N=xx) | 14-Day Vehicle Oil<br>(N=xx) |
|---|---|---|---|---|
| System Organ Class | Not Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Not Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Suspected | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first study drug application.

Note: MedDRA dictionary (Version 20.1)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the strongest reported relationship.



**Statistical Analysis Plan** Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016

Version: 0.03

Date: DD MAY 2019

### 10. INDEX OF PLANNED LISTINGS

| Listing 16.1.7: Randomization Scheme | 81 |
|---|---|
| Listing 16.2.1.1: End of Study Information | 82 |
| Listing 16.2.1.2: Discontinued Subjects | 83 |
| Listing 16.2.1.3: Screen Failures | 84 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations | 85 |
| Listing 16.2.3: Analysis Populations | 86 |
| Listing 16.2.4.1: Subject Demographic Information | 87 |
| Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System Organ Classes and Preferred Terms | 88 |
| Listing 16.2.4.2.2: Medical History | 89 |
| Listing 16.2.4.3: Physical Examination | 90 |
| Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DDE ATC Level 2 Terms and Preferred Names | |
| Listing 16.2.4.3.2: Prior and Concomitant Medications | 92 |
| Listing 16.2.4.4: Prior and Concomitant Procedures/Therapies | 93 |
| Listing 16.2.5.1: Study Visit Compliance | 94 |
| Listing 16.2.5.2: Subject Dosing Compliance | 95 |
| Listing 16.2.5.3: Missed/Extra Doses | 96 |
| Listing 16.2.5.4: Study Drug Dispensing and Return | 97 |
| Listing 16.2.6.1: Otomycosis Signs and Symptoms | 98 |
| Listing 16.2.6.2: Subject Global Assessment | 99 |
| Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms | .100 |
| Listing 16.2.7.2.2: Pre-Treatment Adverse Events | .101 |
| Listing 16.2.7.2.3: Treatment-Emergent Adverse Events | .102 |
| Listing 16.2.7.2.4: Serious Adverse Events | .103 |
| Listing 16.2.8.1.1: Urine Pregnancy Test Results | .104 |
| Listing 16.2.8.2.1: Microbial Culture Results | .105 |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

## Listing 16.1.7: Randomization Scheme (Page xx of yy)

| Subject | Age/Sex | Eval | Randomization Date | Assigned Arm | Treated Ear(s) | Worse Ear |
|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxx xxxxxx | xxxx | xxx xxxxx xxxx xxxx<br>xxxxx xxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxx xxxxxx | xxxxx | |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxx xxxxxx | xxxx | |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016

Version: 0.03 Date: DD MAY 2019

Listing 16.2.1.1: End of Study Information
Treatment Arm
(Page xx of yy)

| Subject | Age/Sex | Eval | Date of<br>First Dose<br>of Study Drug | Date of<br>Last Dose of<br>Study Drug | Reason for<br>End of Treatment | Reason for Study<br>Completion/<br>Discontinuation | Date of Study<br>Completion/<br>Discontinuation<br>(Day) 1 |
|---|---|---|---|---|---|---|---|
| XXXXXX | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | xxxx xx xxxxxxxxx | xxxx xx xxxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxx | xxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx xxxxxxxx x xxx | ********* ******** * *** | xxxxxxxxx xxxx |
| XXXXXX | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.1.2: Discontinued Subjects
Treatment Arm
(Page xx of yy)

| Subject | Age/Sex | Eval | Date of<br>First Dose<br>of Study Drug | Date of<br>Last Dose of<br>Study Drug | Reason for<br>End of Treatment | Reason for Study<br>Completion/<br>Discontinuation | Date of Study<br>Completion/<br>Discontinuation<br>(Day) 1 |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx xxxx |
| xxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx xxxx |
| xxxxx | XXXX | xxxxx | xxxxxxxxx | xxxxxxxxx | xxxx xx xxxxxxxxx | xxxx xx xxxxxxxx | xxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx xxxx |
| xxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |
| xxxxx | xxxx | xxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx xxxxxxxx x xxx | ********* ******** * *** | xxxxxxxxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx xxxx |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

## Listing 16.2.1.3: Screen Failures (Page xx of yy)

| Subject | Age/Sex | Date of<br>Screen Failure | Failed Inclusion<br>Met Exclusion<br>Criteria | n/<br>Criteria | Other Reason for Screen Failure |
|---|---|---|---|---|---|
| xxxxxx | xxxxxxx | xxxxxxxxx | xxx | xxxxxxxx xxxxxxx x | |
| xxxxxx | xxxxxxx | xxxxxxxxx | xx | | xxxx xxx xxx xx xxxxxx |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

## Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations (Page xx of yy)

| Subject | Age/Sex | Eval | Date<br>Assessed | Criteria<br>Failed | Description |
|---|---|---|---|---|---|
| XXXXXX | xxxx | xxxxxxxx | xxxxxxxxx | xxxxx | ***** *** ** ******* **** *********** **** |
| xxxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxxx | ***** *** ** ****** **** **** * ******* |
| xxxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxxx | ***** ** ******* ** ***** *** ** ****** |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


## Listing 16.2.3: Analysis Populations Treatment Arm (Page xx of yy)

Subject Age/Sex Population Included Reason(s) Excluded Exceptions xxxxxx XXXX Intent-to-Treat XXX Modified Intent-to-Treat XXX Per-Protocol XXX Safety XXX Intent-to-Treat XXXXXX XXXX XXX Modified Intent-to-Treat XXXPer-Protocol XX Safety XXXIntent-to-Treat XXXXXX XXXX XXX Modified Intent-to-Treat XXX Per-Protocol XXX Safety XXX Intent-to-Treat XXXXXX XXXX XXX Modified Intent-to-Treat xxx Per-Protocol XXX Safety XXX XXXXXX XXXX Intent-to-Treat XXX Modified Intent-to-Treat XXX Per-Protocol XXXSafety XXX xxxxxx XXXX Intent-to-Treat XXX Modified Intent-to-Treat XXX Safety XXX Per-Protocol XXX



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.4.1: Subject Demographic Information
Treatment Arm
(Page xx of yy)

| Subject | Eval | A: Age<br>S: Sex | R: Race<br>E: Ethnicity | Date of Birth | C: Childbearing Potential B: Method of Contraception | P: Protocol Version I: Informed Consent Date A: Informed Assent Date |
|---|---|---|---|---|---|---|
| xxxxx | xxxxxxxx | A: xx<br>S: xxxx | R: xxxxx<br>E: xxxxxxxx xx<br>xxxxxx | xxxxxxxxx | C: xx<br>B: | P: xxxxxxx x<br>I: xxxxxxxxxx<br>A: xx |
| xxxxx | xxxxxxxx | A: xx<br>S: xxxxxx | R: xxxxxxx<br>E: xxx xxxxxxx<br>xx xxxxxx | xxxxxxxx | C: xxx<br>B: xxxx xxxxxxxx | P: xxxxxxx x<br>I: xxxxxxxxx<br>A: xx |
| xxxxx | xxxxxxxx | A: xx<br>S: xxxx | R: xxxxx<br>E: xxx xxxxxxxx<br>xx xxxxxx | xxxxxxxxx | C: xx<br>B: | P: xxxxxxx x<br>I: xxxxxxxxxx<br>A: xx |

\_\_\_\_\_\_



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Condition or Surgery Verbatim Term |
|---|---|---|
| xxxxx xxx xxxxxxxx xxxxxxx xxxxxxxx | xxxx xxxxxxxxx xxxxxxx | xxxx xxxxxxxxx xxxxxx |
| | xxxxxxxxxxxx | xxxxxxxxxxxx |
| xxxxxxx xxxxxxxx | xxxxxxxxx | xxxxxx xxxxxxxx |
| | xxxxx xxxxxxxxxx | xxxxxx xxxxxxxxx |
| | | xxxxxx xxxxxxxxxxx |
| | *********** | xxx xxxxxx xx xxxxx |
| | xxxxx xxxxx xxxxx xxxxx | xxxxx xxxxxx xxxxxx xxxxx |
| | xxxxxx xxxxxx xxxxxxxx | xxxxxxxxx xxxxx xxxxxxx |
| | xxxxxxxxxxx xxxxxxx | xxxxxxxxxxx xxxxxxx |
| | xxxxxxx xxxxxx xxxxxxx | xxxxxxx xxxxx xxxxxx |
| | xxxxxxxx xxxxxxxxx | xxxxxxxxx xxxxxxx |
| | | xxxxxxxxx xxxxxxxxx |
| | xxxxxxxxx xxxxxxx | xxxxxxxxxx xxxxxxx xxxxxxx xx |
| | xxxxxxxx xxxxx xxxxxxxxxx | xxxx xxxxxxxx xxxxxxxxxxx |
| ********* ******* *** ******* | *************** | ***** ******* ****** ****** |
| | xxxxxxx xxxxxxxx xxxxxxx | xxxxxxxxx |
| xxx xxx xxxxxxxx xxxxxxxxx | xxxxxxx | xxxxxx xxxx |

Note: System Organ Class and Preferred Term from MedDRA Version 20.1.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.4.2.2: Medical History
Treatment Arm
(Page xx of yy)

| Subject | Age/Sex | Eval | Condition or Surgery<br>Verbatim Term | Physical<br>Exam Finding | P: MedDRA Preferred Term<br>S: MedDRA System Organ Class | | Start Date<br>End Date |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxxx | xxxxxx | xxx | P: xxxxxx<br>S: xxxxxxxxxxx xxxxxxxx xxx xxxxxxxxx<br>xxxxxx | S: x<br>E: x | |
| | | | xxxxxx xxxxxx | xx | P: xxxxxxx<br>S: xxxxxxxxx xxx xxxxxxxx xxxxxxxx | | xxxxxx |
| | | | xxxxxxxxxxx | XX | P: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | S: x<br>E: x | xxxxxx |
| | | | xxxxxxxx | xx | | S: x<br>E: x | xxxxx<br>xxxxxx |
| xxxxxx | xxxx | xxxxxxxxx | xxxx xxxxxxxxxx | xxx | P: xxxxx xxxxxxxxx xxxxxxxx<br>S: xxxxxxxxxx | S: x<br>E: x | xxxxxx |
| | | | xxxxxxxx | xx | | S: x<br>E: x | xxxxxx |
| | | | xxxxxxx xxxxxxxx | xx | P: xxxxxxxx xxxxxxx<br>S: xxxxxx xxxxxx xxxxxxxx | S: x<br>E: x | xxxxxx |
| | | | xxxxxxxx | xx | P: xxxxxxxxx<br>S: xxxxxxxx xxx xxxxxxx xxxxxxxxx | S: x<br>E: x | |
| xxxxxx | xxxx | xxxxxxxxx | ************ | xx | P: xxxxxx xxxxxxxx<br>S: xxxxxxx xxx xxxxxxx xxxxxxxxx | S: x<br>E: x | |
| | | | XXXX XXXXXX XXXXXX XXXX | xx | P: xxxxxx xxxx xxxxxxxx<br>S: xxxxxxxxxxxxxx | S: x<br>E: x | |

Note: System Organ Class and Preferred Term from MedDRA Version 20.1. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Verbatim Term, Start Date, and End Date.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

# Listing 16.2.4.3: Physical Examination Treatment Arm (Page xx of yy)

Physical Exam Visit Subject Age/Sex Eval Date Performed XXXXXX XXXX XXXXXXX XXXXXXX XXXXXXXXX XXX xxxxxxxxxx xxxxxxxxx XX XXXXXX XXXX XXXXXXX XXXXXXX XXXXXXXXX XX XXXXXXXXXX XXXXXXXXX XXX XXXXXXXXXX XXXXXXXXX XXX

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


## Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DDE ATC Level 2 Terms and Preferred Names (Page xx of yy)

| | <del></del> | | <del></del> |
|---|---|---|---|
| ATC Level 2 Term | Standardized Medication Name | Medication Name | I: Indication<br>R: Route |
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| xxxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |

Note: Standardized Medication Name and ATC Level 2 Term map to the WHO-DDE (Version March 1, 2017).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Standardized Medication Name, Medication Name, Indication, and Route.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.4.3.2: Prior and Concomitant Medications Treatment Arm (Page xx of yy)

D: Dose S: Subject M: Medication Name P: Standardized F: Date of First Dose U: Units A: Age/Sex I: Indication Medication Name S: Start Date (Day) 1 F: Frequency E: Eval A: Applied at Dosing Site A: ATC Level 2 Term E: End Date (Day) 1 O: Route S: xxxxxx M: xxxxxxxxxxxx P: xxxxxxxxxxxxx F: xxxxxxxxxx D: xx U: xx A: xxxx I: XXXXXXXX A: xxxxxxxxxxxxx S: xxxxxxxxxx F: xxxx E: xxxxxxxxx A: xx E: xxxxxxx O: xxxxxx M: xxxxxxxxxxxx P: xxxxxxxxxxxxx F: xxxxxxxxxx D: xxxxx I: xxxxxxxx S: xxxxxxxxxx U: xx A: xxxxxxxxxxxx A: xxx E: xxxxxxx F: xx O: xxxx S: xxxxxx M: xxxxxxxxxxxx P: xxxxxxxxxxxxx F: xxxxxxxxxx D: xxx A: xxxx I: XXXXXXXX A: xxxxxxxxxxxx S: xxxxxxxxxx U: xx A: xx E: xxxxxxx F: xx E: xxxxxxxxx O: xxxx

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: Standardized Medication Name and ATC Level 2 Term map to the WHO-DDE (Version March 1, 2017).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

## Listing 16.2.4.4: Prior and Concomitant Procedures/Therapies Treatment Arm (Page xx of yy)

Procedure/ Applied at S: Start Date (Day) 1 Subject Age/Sex Eval Date of First Dose Dosing Site E: End Date (Day) 1 Theraphy Indication XXXX xxxxxxxxx xxxxxxxxxxxx xxxxxxx S: xxxxxxxxx xxxx XXXXXX XXXXXXXX XX E: xxxxxxx XXXXXXXXXXXX XXXXXXX XXX S: xxxxxxxxx xxxx E: xxxxxxx xxxx S: xxxxxxxxx xxxx XXXXXX XXXX XXXXXXXX XXXXXXXXX XXXXXXXXXXXX XXXXXXX XX E: xxxxxxx xxxx

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.5.1: Study Visit Compliance
Treatment Arm
(Page xx of yy)

Study Within Visit Not Done/ Ear(s) Subject Age/Sex Eval Visit Day¹ Visit Window Reason for Unscheduled Visit Cleaned Visit Date XXXXXX XXXX XXXXXXXX XXXXXXXX XXXXXXXXX XX XXX XXXXX XXXXXX XXXXXXXX XXXXXXXXX XX XXX XXXX XXXXXX XXXXXXXXX XXXXX XXXX XXXXXX XXXX XXXXXXX XXXXXXXX XXXXXXXXX XX XXX XXXXXX XXXXX xxxxxxx XXXXXXXXX XXX XXXX XX XXXXXX XXXXXXXXX XX XXX XXXXX xxxxxxxxx XXXXXX XX XXX XXXXX

Day is calculated as date - baseline date for dates prior to baseline visit. Otherwise, day is calculated as date - Baseline date + 1 for dates on or after baseline visit.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

## Listing 16.2.5.2: Subject Dosing Compliance Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | F: Date of First Dose L: Date of Last Dose | Number<br>of Days<br>of<br>Exposure | Calculated <sup>1</sup> Number of Applications | Amount<br>of Study<br>Drug<br>Used (g) | Percent<br>Compliant | Compliant? <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxx | XX | xx | xxxx | XXX | xxx |
| xxxxx | xxxx | xxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxx | xx | xx | xxxx | xxx | xxx |
| xxxxxx | xxxx | xxxxxxxx | F: xxxxxxxxxx<br>L: xxxxxxxxxx | xx | XX | xxxx | xxx | xxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing Format May Be Altered on Confirmation of Dosing Data Capture.

The number of applications will be calculated by 2\*(Date of Last Dose - Date of First Dose + 1) - (Number of Doses Missed) + (Number of Extra Doses).

<sup>&</sup>lt;sup>2</sup> A subject was considered compliant with the dosing regimen if the subject applied 80% to 120% of the total number of expected doses during the treatment period.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.5.3: Missed/Extra Doses
Treatment Arm
(Page xx of yy)

| Subject | Age/Sex | Eval | Date of First Dose | Treatment<br>Ear(s) | Date of Missed/<br>Extra Dose | Number of<br>Missed Doses | Number of<br>Extra Doses |
|---|---|---|---|---|---|---|---|
| xxxxx | XXXX | xxxxxxxx | xxxxxxxx | xxxx | xxxxxxxxx | х | |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxxx<br>xxxx | xxxxxxxxx<br>xxxxxxxxx | x | х |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxx | xxxxxxxxx | х | |
| | | | | XXXX | XXXXXXXXX | Х | X |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

# Listing 16.2.5.4: Study Drug Dispensing and Return Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Kit<br>Number | Bottle<br>Number | Date<br>Dispensed | Dispense<br>Weight | Return<br>Date | Return<br>Weight |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxx | х | xxxxxxxxx | xxx | xxxxxxxxx | xxx xxxx |
| xxxxxx | XXXX | xxxxxxxx | xxxxx | Х | xxxxxxxxx | xxxxx | xxxxxxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxxx | XXXXX | Х | xxxxxxxxx | xxxxx | xxxxxxxxx | xxxxx |
| xxxxxx | XXXX | xxxxxxxx | xxxxx | Х | xxxxxxxxx | xxxxx | xxxxxxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | Х | xxxxxxxx | xxxxx | xxxxxxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | Х | xxxxxxxx | xxx | xxxxxxxxx | xxx xxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | Х | xxxxxxxx | xxxxx | xxxxxxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | Х | xxxxxxxxx | xxxxx | xxxxxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | Х | xxxxxxxx | xxxxx | xxxxxxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | Х | xxxxxxxxx | xxxxx | xxxxxxxxx | xxxxxx |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


| S: Subject<br>A: Age/Sex<br>E: Eval | V: Visit<br>D: Date | Assesor | Investigator<br>Initals | Ear | Pruritus | Debris | Presence of<br>Fungal Elements | Pain |
|---|---|---|---|---|---|---|---|---|
| S: xxxxx<br>A: xxx<br>E: xxxxxxx | V: xxxxxxxxx<br>D: xxxxxxxxxx | xxxxxx | | xxxx | xxxxxxx | | | |
| I. MAMMAMA | V: xxx xx<br>D: xxxxxxxxx | xxxxxxxxxx | xxx | XXXX | xxxxxxx | xxxxxxx | xxxxx | xxxxxxx |
| | V: xxx xx<br>D: xxxxxxxxx | xxxxxxxxxx | xxx | xxxx | xxxxxxx | xxxxxxx | xxxxx | xxxxxxx |
| S: xxxxx<br>A: xxxx | V: xxxxxxxxx<br>D: xxxxxxxxx | xxxxxx | | xxxx | xxxxxxx | | | |
| E: xxxxxxxx | V: xxx xx<br>D: xxxxxxxxx | xxxxxxxxxx | xxx | xxxx | xxxxxxx | xxxxxxx | xxxxxx | xxxxxxx |
| | V: xxx xx<br>D: xxxxxxxxx | xxxxxxxxxx | xxx | xxxx | xxxxxxx | xxxxxxx | xxxxx | xxxxxxx |

\_\_\_\_\_



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.6.2: Subject Global Assessment Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Date | Visit | Ear | Subject Global Assessment |
|---|---|---|---|---|---|---|
| «xxxx | xxxxx | xxxxxxxxxxx | xxxxxxxxx | xxxxxxx | xxxx | x x xxxxxxxx |
| | | | | | XXXXX | x x xxxxxxxx |
| | | | xxxxxxxxx | XXXXXXX | XXXX | x x xxxxxxxx |
| | | | | | XXXXX | x x xxxxxxxx |
| | | | XXXXXXXXX | XXX XX | XXXX | x x xxxxxxxx |
| | | | | | XXXXX | x x xxxxxxxx |
| | | | XXXXXXXXX | XXX XX | XXXX | X X XXXXXXX |
| | | | | | XXXXX | x x xxxxxxxx |
| XXXXX | XXXXX | XXXXXXXXXXX | xxxxxxxxx | xxxxxxx | XXXX | x x xxxxxxxx |
| | | | | | XXXXX | x x xxxxxxxx |
| | | | XXXXXXXXX | XXXXXXXX | XXXX | X X XXXXXXXX |
| | | | | | XXXXX | X X XXXXXXX |
| | | | XXXXXXXXX | XXX XX | XXXX | X X XXXXXXX |
| | | | | | XXXXX | x x xxxxxxxx |
| | | | XXXXXXXXX | XXX XX | XXXX | x x xxxxxxxx |
| | | | | | XXXXX | X X XXXXXXX |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Adverse Event |
|---|---|---|
| xxxxx xxxxx xxxxx | xxxxx xxxxx xxxxx | xxxxxxxxx |
| | | xxxxxxx xxxxxxx xxxxxxxx |
| | | ******** ******** ********** |
| | xxxxx xxxxx xxxxx | XXXXXXXXX |
| | AAAAA AAAAA | ******** ********* |
| | | ******** |
| | xxxxxxxxx | xxxxx xxxxx xxxxx |
| | | xxxxxxx xxxxxxx xxxxxxxxx |
| | | xxxxxxx xxxxxxxx xxxxxxxxxxxx |

Note: System Organ Class and Preferred Term map to MedDRA (Version 20.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, Preferred Term, and Adverse Event.



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

## Listing 16.2.7.2.2: Pre-Treatment Adverse Events Treatment Arm (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | A: Adverse Event Description C: System Organ Class P: Preferred Term | F: Date of First Dose S: Start Date (Day) 1 E: End Date (Day) 1 B: When Did The AE Begin | E: Occur on the Ear D: Occur at Dosing Site S: Severity R: Relationship to Study Drug O: Outcome | S: Serious<br>A: Action Taken<br>T: Other Action<br>D: Cause Discontinuation |
|---|---|---|---|---|
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxxxxxxx | E: xxxxxxx xxx xxx xxx xx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxxxxxxxx | XX XXX XXXX | A: xxxx xxx xxxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx | D: xx | T: xxxxxxxxxx xxxxx xxxxx |
| | | B: xxxxxxxxxx xxxxx | S: xxxxxxxx | D: xx |
| | | XXXX XX XXXXX XXXX | R: xxx xxxxxxxx | |
| | | | O: xxxxxxxxxxxxxxxx | |
| | | | XXXX XXXXXXX | |

Note: System Organ Class and Preferred Term map to MedDRA (Version 20.1).

Listing sorted by Subject, Start Date, End Date, and Adverse Event Description.

¹ Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

# Listing 16.2.7.2.3: Treatment-Emergent Adverse Events Treatment Arm (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | A: Adverse Event Description C: System Organ Class P: Preferred Term | F: Date of First Dose S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> B: When Did The AE Begin | E: Occur on the Ear D: Occur at Dosing Site S: Severity R: Relationship to Study Drug O: Outcome | S: Serious A: Action Taken T: Other Action D: Cause Discontinuation |
|---|---|---|---|---|
| S: xxxxxx | A: xxxxxxxxxxxx | F: xxxxxxxxx | E: xxxxxxx xxx xxx xxx xx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxxxxxxx | xx xxx xxxx | A: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxxxxxxx | D: xx | T: xxxxxxxxxx xxxxx xxxxx |
| | | B: xxxxxxxxxx xxxxx | S: xxxxxxxx | D: xx |
| | | XXXX XX XXXXX XXXX | R: xxx xxxxxxxx | |
| | | | O: xxxxxxxxxxxxxxxx | |
| | | | XXXX XXXXXXX | |

Note: System Organ Class and Preferred Term map to MedDRA (Version 20.1).

Listing sorted by Subject, Start Date, End Date, and Adverse Event Description.

¹ Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

## Listing 16.2.7.2.4: Serious Adverse Events Treatment Arm (Page xx of yy)

| Description<br>System Organ Class | F: Date of First Dose<br>S: Start Date (Day) <sup>1</sup><br>E: End Date (Day) <sup>1</sup><br>B: When Did The AE Begin | D: Occur at Dosing Site S: Severity R: Relationship to Study Drug O: Outcome | S: Serious A: Action Taken T: Other Action D: Cause Discontinuation |
|---|---|---|---|
| xxxxxxxxxxxx | F: xxxxxxxxxx<br>S: xxxxxxxxxx<br>E: xxxxxxxxxxx<br>B: xxxxxxxxxxx xxxx | E: xxxxxxxx xxx xxx xxxx xx<br>xx xxx xxxx<br>D: xx<br>S: xxxxxxxx<br>R: xxx xxxxxxxxx | S: xxx A: xxxx xxx xxxxxxx T: xxxxxxxxxxx xxxxx xxxxx D: xx |
| | Adverse Event Description System Organ Class Preferred Term *********************************** | Description S: Start Date (Day)¹ System Organ Class E: End Date (Day)¹ Preferred Term B: When Did The AE Begin xxxxxxxxxxxxxxx F: xxxxxxxxx xxxxxxxxxx | Adverse Event F: Date of First Dose S: Severity Description S: Start Date (Day) 1 R: Relationship to System Organ Class E: End Date (Day) 1 Study Drug Preferred Term B: When Did The AE Begin O: Outcome ***XXXXXXXXXXXXX F: XXXXXXXX |

Note: System Organ Class and Preferred Term map to MedDRA (Version 20.1).

Listing sorted by Subject, Start Date, End Date, and Adverse Event Description.

¹ Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


Date: DD MAY 2019

#### 

| Subject | Age/Sex | Eval | Visit | Date | Results |
|---------|---------|----------|--------------|-----------|----------|
| XXXXXX | XXXX | XXXXXXXX | xxxxxxxx | xxxxxxxxx | XXXXXXX |
| | | | XXXXXXXX | XXXXXXXXX | XXXXXXXX |
| | | | XXXXXX | XXXXXXXXX | XXXXXXXX |
| | | | XXXXXX | XXXXXXXXX | XXX XXXX |
| | | | XXXXXX | XXXXXXXXX | XXXXXXX |
| | | | XXXXXXXXXXXX | XXXXXXXXX | XXXXXXXX |
| XXXXXX | XXXX | XXXXXXXX | XXXXXXXX | XXXXXXXXX | XXXXXXXX |
| | | | XXXXXXX | XXXXXXXXX | XXXXXXXX |
| | | | XXXXXX | XXXXXXXXX | XXXXXXXX |
| | | | XXXXXX | XXXXXXXXX | XXXXXXX |
| | | | XXXXXX | XXXXXXXXX | XXXXXXX |
| | | | xxxxxxxxxxxx | xxxxxxxxx | xxxxxxx |



Hill Dermaceuticals, Inc. HD-MCZ-PHII-DRF062016


(Page xx of yy)

| Subject | Age/Sex | Eval | Ear | Date | Visit | Culture Type | Results |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxxx | xxxxx | ****** | xxxxxxxx<br>xxx xx xxxxxxxxx | xxxxxx<br>xxxxxxx | xxxxx xxxxxxx xxxx<br>xx xxxxx xxxxxxxx |
| xxxxx | xxxx | xxxxxxxx | xxxxx | ********* | ************************************** | XXXXXXXX<br>XXXXXXXX<br>XXXXXXX | ***** ****** **** ***** ***** ****** **** ***** ** ***** ****** |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, Category, and Lab Test.